CLINICAL TRIAL: NCT01140321
Title: A Randomized, Open-label Therapeutic Trial Evaluating the Efficacy and Safety of Neridronate (Nerixia®) in the Treatment of Osteoporosis in Patients With Thalassemia Major and Severe Thalassemia Intermedia.
Brief Title: Efficacy and Safety of Neridronate (Nerixia®)to Treat Osteoporosis in Patients With TM and TI
Acronym: Nerixia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Collaborators: Ospedale Maggiore Policlinico Mangiagalli e Regina Elena (Other); Ospedale "Perrino" Brindisi (Unknown); Reggio Calabria (Other); Azienda Ospedaliera Villa Sofia (Unknown); Azienda Ospedaliera V. Cervello (Other); Università di Ferrara (Unknown); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Dr. Gian Luca Forni, MD, Ente Ospedaliero Ospedali Galliera
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60/2003/Nerixia
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Osteoporosis; Thalassemia Major; Thalassemia Intermedia
Keywords: Thalassemia; Neridronate; Osteopenia; Osteoporosis
MeSH Terms: conditions — Osteoporosis; beta-Thalassemia; Thalassemia; Bone Diseases, Metabolic | interventions — 6-amino-1-hydroxyhexane-1,1-diphosphonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neridronato (Experimental): Thalassemia Major or Severe Thalassemia Intermedia
  Interventions: Drug: Neridronate
- Placebo (No Intervention): Thalassemia Major or Severe Thalassemia Intermedia

INTERVENTIONS:
Drug: Neridronate — Neridronate is an aminobisphosfonate of third generation that has been proved in several clinical trials to have the ability to inhibit osteoclast-mediated bone resorption and it is generally well tollerated also at high doses. Thanks to these properties it has been used in the treatment of several bone disorders such as Paget's disease and Osteogenesis Imperfecta. Neridronate, given intravenously or orally (tablets), reduces both the levels of bone alcaline phosphatase and of the other markers of bone resorption activity. Recently it has been approved by the Italian Ministry of Health for the commercialization with the indication "Osteogenesis Imperfecta".
  Arms: Neridronato

SUMMARY:
An Italian Multicentric randomized, open-label therapeutic trial evaluating the efficacy and safety of Neridronate in the treatment of Osteoporosis in patients with Thalassemia Major and Severe Thalassemia Intermedia.

Efficacy and safety of the drug will be evaluated measuring at every visit this parameters:

* haematological: Haemochrome
* blood chemistry: creatinine, BUN, AST, ALT, Ca, P, proteins electrophoresis, total proteins.

The prevalence of ectopic calcification and pseudoxantoma elasticum (PXE)-like syndrome and their follow-up will be evaluated at the beginning of the study vs 24 months through physical examination, abdominal echography and fundus oculi examination.

During the trial other known risks factors for osteoporosis will be recorded, including prevalence and incidence of bone fractures and, if executed, Polimorphisms COLIA1.

At the beginning of the study and at months 12 and 24 morphometry DXA will be performed to evaluate of the presence of bone deformities.

Furthermore data regarding QOL and symptom pain will be evaluated trough administration of scale SF-36.

At 12 months an intratrial analisis will be performed on efficacy and safety parameters in order to introduce possible amendments to the study design and to decide the prosecution of the trial

During the trial all adverse events will be recorded

DETAILED DESCRIPTION:
Aim of the Study At present, due to the global therapeutic approach, the prognosis of Thalassemia Major and Severe Thalassemia Intermedia is open-ended. Regular transfusional regimens from childhood and early iron chelation therapy prevent bone deformities that in the past characterized this disease even though according to several authors a high percentage of patients suffers from osteopenia-osteoporosis. This persistent complication may be explained by one or more coexistent factors such as anaemia, genetic factors, sex hormones involved in the bone metabolism, iron and chelation therapy, hypothiroidism, low or subnormal concentrations of serum vitamin D, etc.

Pain resulted to be the only parameter that may be considered to distinguish patients with Thalassemia Major from healthy patients of the same age through a survey about Quality of Life performed in the Center of Genoa. More frequently pain is localized in the lumbar vertebrae, it is often described with invalidant pictures and it has to be referred to osteoporosis of vertebral bodies.

The incidence of spontaneous fractures observed in the specialistic centers treating these pathologies is increasing.

Thalassemia Intermedia is an eterogeneous clinical entity including a wide range of phenotypes from mild to severe forms. In the mild forms hemoglobin levels range between 8-9 g/dl, which is stable without the need for regular transfusion therapy unless an intercurrent episode aggravates anemia; no expansion of the bone marrow is observed. By contrast, there are forms in which anemia is persistently more severe (6.5- 7.5 g/dl) with marked ineffective erythropoiesis. In these cases, especially when the diagnosis is made in childhood, patients should receive a transfusional regimen similar to Major forms with similar complications such as osteoporosis.

For these reasons in patients affected with Severe Thalassemia Intermedia and with Thalassemia Major prevention and early diagnosis of osteoporosis are important as well as treatment of the established disease in order both to improve quality of life and life expectancy.

In therapeutical trials previously described bisphosphonates have been shown to be effective because of their ability to inhibit bone resorption and their relatively few side effects resulting in an increase bone density. Since all the previous trials were conducted on a small number of patients, we propose a randomized, open label large multicentric trial to test the efficacy of Neridronate. The possibility to administrate this drug every 90 days intravenous makes dosing regimens simple and reduces the frequency of administration. These are important factors to improve adherence to therapy in patients already subjected to an heavy daily therapeutic load.

Primary Objectives The primary objective of this study is to evaluate the efficacy of Neridronate (an aminobisphosfonate of third generation that has been proved in several clinical trials to have the ability to inhibit osteoclast-mediated bone resorption) to increase Bone Mass Density (BMD) measured through Double X-ray densitometry (DXA). Bone densitometry will be performed at basal screening and then at 6, 12, 18, 24 months from the beginning of the treatment.

Secondary objectives The effect of Neridronate on bone turn over will be evaluated through bone alcaline phosphatase (BALP) and telopeptide C-terminal of type 1 seric collagen (CTX-s), at screening and then at 6, 12, 18, 24 months from the beginning of the treatment.

The dosage of the markers will be centralized. Study design An Italian Multicentric randomized, open-label therapeutic trial evaluating the efficacy and safety of Neridronate in the treatment of Osteoporosis in patients with Thalassemia Major and Severe Thalassemia Intermedia.

Efficacy and safety of the drug will be evaluated measuring at every visit this parameters:

* haematological: Haemochrome
* blood chemistry: creatinine, BUN, AST, ALT, Ca, P, proteins electrophoresis, total proteins.

The prevalence of ectopic calcification and pseudoxantoma elasticum (PXE)-like syndrome and their follow-up will be evaluated at the beginning of the study vs 24 months through physical examination, abdominal echography and fundus oculi examination.

During the trial other known risks factors for osteoporosis will be recorded, including prevalence and incidence of bone fractures and, if executed, Polimorphisms COLIA1 At the beginning of the study and at months 12 and 24 morphometry DXA for the evaluation of the presence of bone deformities Furthermore data regarding QOL and symptom pain will be evaluated trough administration of scale SF-36.

During the trial all adverse events will be recorded

Extension study:

Objectives of the extension study

1. In vitro analysis of the effects of iron overload and chelating molecules on mesenchymal stem cells growth and osteogenic differentiation
2. Evaluation of the effects of neridronate on normal and thalassemic MSCs'proliferation and differentiation.
3. Phenotypical characterization of MSCs prepared from thalassemic patients treated with or without neridronate Study design A. In vitro analysis of the effects of iron overload and chelating molecules on MSCs growth and osteogenic differentiation B. Evaluation of the effects of neridronate on normal and thalassemic MSCs'proliferation and differentiation.

C. Phenotypical characterization of MSCs prepared from thalassemic patients treated with or without neridronate A. In vitro analysis of the effects of iron overload and chelating molecules on MSCs growth and osteogenic differentiation

1. Preparation of a collection of bone marrow mesenchymal stem cells from normal subjects To isolate and prepare MSCs, we will utilize the protocol described in detail in Oliva et. al. (Molec. and Cell. Biochem., 2003, 247:55-60). The details of MSCs preparation are reported in annexes.

   The cells expressed specific surface markers, such as CD13, CD29, CD44, CD105, CD166, and were negative for hematopoietic cell markers CD14, CD34 and CD45.

   In this way, we are preparing a normal MSCs'bank, on which perform the experimentation. At present, we have already available more than 10 preparations of MSCs from normal subjects.
2. Analysis of the effects of iron overload on proliferation and differentiation of MSCs Although it is well known that thalassemic subjects undergo iron overload, no data are available in Literature on the effects of this metal on proliferation and differentiation of MSCs. To this aim we will proceed as indicated below. We will evaluate the proliferation rate and iron and ferritin intracellular levels in MSCs in logarithmic phase incubated with increasing concentrations of iron, starting from physiological hematic amounts, i.e. 2-18 microg/ml, until reaching values 10-fold higher, similar to those occurring in thalassemic patients. We will analyze the effect on growth rate by direct cell count, MTT vitality assay, and 3H-thymidine incorporation (DNA synthesis).

   Successively we will analyze the effects of iron overload on the levels of the main proteic product of MSCs, namely type I collagen, following the protocol reported. Confluent cultures of early passages (0-3) of MSCs, nontreated and treated with iron overload, are tripsinized, counted and centrifuged at 800xg. The pellets are resuspended in 0.5 M acetic acid containing 250 microg/ml pepsin.

   After 16 hours of gentle shaking at 4°C, the insoluble residue is pelleted at 20.000xg for 1 hour, solubilized in run buffer and analyzed by 6% SDS-PAGE. Afterwards, proteins are blotted to a nitrocellulose membrane and incubated with rabbit monoclonal antibodies specific for human type I collagen. The immunoreactive bands are then incubated with horse radish peroxidase conjugated secondary antibodies and detected by means of enhanced chemoluminescent technique (ECL).

   The effects on differentiation will be evaluated analyzing the expression of specific markers of osteoblastic phenotype, namely alkaline phosphatase activity and osteocalcin production. In addition, we will evaluate the osteogenic capacity of MSCs expressed by extracellular matrix mineralization. Confluent cultures are incubated with an osteogenic medium composed of dexametasone 100 nM and beta-glycerophosphate 10 mM. If osteogenic capacity is present, calcification noduli appear within 2-4 weeks. To further confirm the matrix mineralization we will measure calcium levels and finally carry out a specific stain by von Kossa method.
3. Analysis of effects of iron chelating molecules on proliferation and differentiation of MSCs We will evaluate the effects of DFO, which represents so far the most used chelating molecule in the therapy of thalassemia in spite of the well known disadvantages and toxicity. MSCs cultures, nontreated or treated with iron overload, will be added with DFO at concentrations similar to those obtained in vivo following drug administration to thalassemic patients. We will analyze the effect of the treatment on growth rate, collagen type I levels, alkaline phosphatase activity, osteocalcin production, as well as the osteogenic capacity.
4. Characterization of cell cycle components in MSCs subjected to iron overload and/or DFO It is well known that characterization of cell cycle components represents the basis for the comprehension of pivotal events of proliferation and differentiation processes.

Thus, cell extracts obtained from both MSCs cell populations treated as described above (i.e. iron, DFO or iron overload and/or desferrioxamine) will be analyzed by immunoblotting employing antibodies against several cycle proteic components. Among them in particular: cyclin D1, D2, and D3, cyclin E, cyclin A; CDK4, CDK6, CDK2 and CDK1; p16, p14, p15, p21, and p27. Moreover, the phosphorylation of the retinoblastoma protein and the cdk activities will be analyzed.

B. Evaluation of the effects of neridronate on normal and thalassemic MSCs'proliferation and differentiation.

The objective of this study will be the in vitro analysis of the effects of the neridronate on normal and thalassemic human MSCs. In particular, we will evaluate if the drug, tested at concentrations between 10(-4) M and 10(-6) M being 10(-5) M the therapeutic dose, affect the viability, proliferation, and cellular activity of MSCs. The effects on proliferation will be assessed in terms of 3H-thymidine incorporation, MTT test and cell cycle engine modulation. The action on differentiation will be evaluated analyzing the expression of specific markers, namely type I collagen levels, alkaline phosphatase activity and osteocalcin production. In addition, we will evaluate the osteogenic capacity of MSCs expressed by extracellular matrix mineralization, by the measure of calcium levels and by von Kossa staining.

C. Phenotypical characterization of MSCs prepared from thalassemic patients treated with or without neridronate The aim of this study will be to investigate whether the treatment of thalassemic patients with neridronate might positively affect the osteoporotic condition and, at the same time, improve the osteogenic capacity of MSCs. Therefore, we will prepare MSCs from thalassemic patients treated or not with neridronate and cultivate them according to standard method. In particular, we will analyze the growth rate, the cell cycle machinery, the collagen levels, the AP activity and the osteocalcin synthesis. Most importantly we will evaluate the extracellular matrix mineralization.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting BMD Z score <-2 at the level of the femoral neck or of the lumbar column Regular transfusional regimen in order to mantain pre-transfusional Hb values >9 g/dl.

Written informed consent by the patient

Exclusion Criteria:

Entravenous administration of bisphosphonates within the past 2 years

Administration of di bisphosphonates per os, unless wash out as it follows:

1 year if >8 weeks <48 weeks 6 months if > 2 weeks and <8 weeks Hypoparathyroidism Thalassemia Intermedia if not regularly transfused Pregnancy and breast feeding Impaired renal function (creat. > 1.5 mg/dl) Neoplastic disease Patients with mean levels of alanine aminotransferase ALT > 300 U/l and patients with variations of AST or AST of 300% within the year before randomization. (At least 4 misurations over 12 months) Systemic cardiovascular, renal, hepatic disease etc. which would prevent the patient from undergoing study treatment Known hypersensibility to bisphosphonates. History of non compliance to medical regimens and patients who are considered potentially unreliable and/or not cooperative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gian Luca Forni, MD, Principal Investigator — Centro della Microcitemia e delle Anemie Congenite E.O. Ospedali Galliera- Genova Italy; Ernesto Palummeri, MD, Principal Investigator — S.C. Geriatria E.O. Ospedali Galliera - Genova Italy
Locations (8):
- Italy (8):
  - Divisione di Ematologia, Ospedale "Perrino", Brindisi
  - Dipartimento di Medicina Clinica e Sperimentale, Sezione di Pediatria, Università di Ferrara, Ferrara
  - Centro della Microcitemia e delle Anemie Congenite - Ematologia E.O. Ospedali Galliera, Genova
  - SC Geriatria E.O. Ospedali Galliera, Genova
  - Centro Anemie Congenite, Ospedale Maggiore Policlinico, IRCCS, University of Milan, Milan
  - U.O. "Ematologia II con Talassemia" A.O. " V. Cervello, Palermo
  - U.O. Pediatria II, A.O. "Villa Sofia", Palermo
  - Centro Microcitemia, A.O. B.M.M., Reggio Calabria

REFERENCES:
- [Derived] Forni GL, Perrotta S, Giusti A, Quarta G, Pitrolo L, Cappellini MD, D'Ascola DG, Borgna Pignatti C, Rigano P, Filosa A, Iolascon G, Nobili B, Baldini M, Rosa A, Pinto V, Palummeri E. Neridronate improves bone mineral density and reduces back pain in beta-thalassaemia patients with osteoporosis: results from a phase 2, randomized, parallel-arm, open-label study. Br J Haematol. 2012 Jul;158(2):274-282. doi: 10.1111/j.1365-2141.2012.09152.x. Epub 2012 May 10. PMID 22571408